CLINICAL TRIAL: NCT00537732
Title: Omeprazole and Reflux Disease - Improvement of Clinical Outcome by Genotype-adjusted Dosing
Acronym: GERD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment problems
Sponsor: Matthias Schwab (Other)
Responsible Party: Sponsor-Investigator, Matthias Schwab, MD, Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF)
Organization: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IKP-219; 2006-004650-24 (EudraCT Number)
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Gastroesophageal Reflux
Keywords: gastro-oesophageal reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Active Comparator): 3 tablets, only 20 mg omeprazole, genotype independent
  Interventions: Drug: omeprazole
- intervention group (Active Comparator): 20 vs. 60 mg daily, genotype dependent
  Interventions: Drug: omeprazole

INTERVENTIONS:
Drug: omeprazole — 20 mg daily
  Arms: control group
Drug: omeprazole — 20 vs. 60 mg daily, genotype dependent
  Arms: intervention group

SUMMARY:
Patients with gastroesophageal reflux disease (GERD) are either treated for 4 weeks with a standard dose (20mg) of omeprazole, a drug of first choice, or by an individualized dosing (20 or 60mg/day) according how fast the patient can metabolize (eliminate) the drug. The individual elimination capacity is genetically controlled and therefore all patients will be genotyped prior to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with GERD grade A and B (mild to moderate severe disease) diagnosed by routine endoscopy will be recruited in different clinical and ambulant centres of gastroenterology; written informed consent is obligatory
* Range of Age: 20-70
* BMI: 20-30

Exclusion Criteria:

* Patients who are allergic to proton-pump inhibitors or show incompatibility
* Patients who have lactase deficiency
* Patients who have severe chronic disease
* Patients who participated in another study during the last three months
* Patients who are pregnant

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
endoscopic healing rate in patients with GERD after 4 weeks of individualised dosing of omeprazole (according to metabolic capacity of the patient) | 4 weeks

SECONDARY OUTCOMES:
clinical healing rate in patients with GERD after 4 weeks of individualised dosing of omeprazole | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Schwab, Prof, MD, Principal Investigator — Dr. Margarete Fischer-Bosch-Institute of Clinical Pharmacology
Locations (1):
- Dr. Margarete Fischer-Bosch-Institute of Clinical Pharmacology, Stuttgart, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Klotz U, Schwab M, Treiber G. CYP2C19 polymorphism and proton pump inhibitors. Basic Clin Pharmacol Toxicol. 2004 Jul;95(1):2-8. doi: 10.1111/j.1600-0773.2004.pto950102.x. PMID 15245569